CLINICAL TRIAL: NCT03461055
Title: Lavender Aromatherapy vs Placebo to Decrease Anxiety and Pain During Intrauterine Insemination (IUI).
Brief Title: Lavender During Intrauterine Insemination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elizabeth A. Stewart, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-001147
Record Dates: First submitted 2018-03-05; First posted 2018-03-09 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Infertility, Female; Anxiety
MeSH Terms: conditions — Infertility, Female; Anxiety Disorders | interventions — lavender oil; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender (Experimental): Lavandula angustifolia aromatherapy. 1 drop on a cotton ball placed in a porous pouch. Given to patients at the time of their intrauterine insemination.
  Interventions: Other: Lavender
- Water (Placebo Comparator): 1 drop of water on a cotton ball placed in a porous pouch. Given to patients at the time of their intrauterine insemination.
  Interventions: Other: Water

INTERVENTIONS:
Other: Lavender — Lavender aromatherapy
  Other Names: Lavandula angustifolia
  Arms: Lavender
Other: Water — Water
  Arms: Water

SUMMARY:
The Researchers hope to learn if by using lavender aromatherapy during an intrauterine insemination patients have decreased anxiety and pain at the time of the procedure.

DETAILED DESCRIPTION:
Infertility patients have a high level of anxiety before and during infertility treatments due to anticipated discomfort of a procedure and anticipation of a long awaited pregnancy. Aromatherapy with lavender, an essential oil, has been shown to be effective in reducing anxiety and pain in a variety of procedures such as Botox injections, cesarean delivery and intrauterine device placement.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing intrauterine insemination
* English speaking

Exclusion Criteria:

* Allergy to lavender oil or its components
* Currently using aromatherapy
* Contraindication to intrauterine insemination
* Contraindication to pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Anxiety | During intrauterine insemination procedure
  Anxiety level using a standard visual analog scale. Scale is from 0-100 mm. 0 is absent anxiety. 100 mm is maximal anxiety.

SECONDARY OUTCOMES:
Pain | During intrauterine insemination procedure
  Pain score using Wong-Baker pain scale of 0-10. 0 being absent pain and 10 being maximal pain.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stewart, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States